CLINICAL TRIAL: NCT01205945
Title: The Effect of Abdominal Aortic Aneurysm Screening on Mortality in Asian: A Randomized, Controlled Trial
Brief Title: The Effect of Abdominal Aortic Aneurysm Screening on Mortality in Asian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Jin Hyun Joh, Kyung Hee University East-West Neo Medical Center
Other Study IDs: KHNMC IRB 2010-019
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Aortic aneurysm, abdominal; Screening; Mortality
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Abdominal aortic aneurysm(AAA) occurs when the infrarenal aorta expands to a maximal diameter of 3.0cm or greater. Although AAA may asymptomatic for many years, almost one third eventually rupture if left untreated.

Several randomized trials showed that ultrasonographic screening for AAA could reduce the frequency of acute operations and AAA-related mortality.

However, all of randomized trials were performed in Western countries. There was no randomized trials for AAA screening in Asian countries.

This randomized, controlled trial is to analyze the benefits of screening old population for AAA in Korea.

DETAILED DESCRIPTION:
Old population, aged from 60 to 85 years, are randomized into two groups; one group is invited for ultrasonographic screening for AAA, and the other acts as age- and sex-matched controls.

For screening group, The anterioposterior and transverse diameter of the infrarenal aorta is measured at their maximal sizes. The subsequent surveillance of screened patients is done as follows

* Aortic diameter less than 3.0cm, no further testing
* AAA 3 to 4cm, ultrasonographic follow-up every year
* AAA 4 to 5cm, ultrasonographic follow-up every 6 months
* AAA greater than 5cm, referral to a vascular surgeon

For control group, the information for any causes of death is collected every year.

ELIGIBILITY:
Inclusion Criteria:

* all men aged 60 to 85 years
* women aged 60 to 85 years with cardiovascular risk factors such as hypertension, hyperlipidemia, peripheral arterial occlusive disease, coronary artery disease, cerebrovascular attack.
* men and women older than 50 years with a family history of AAA

Exclusion Criteria:

* people who was diagnosed with AAA
* people who underwent aneurysm repair such as open aneurysm repair or endovascular aneurysm repair
* People who underwent abdominal aortic surgery such as aortobifemoral bypass
* People whose life expectancy is less than 2 years
* People who appear unfit for repair of AAA
* people who do not agree with this study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Popultaion who reside in Korea as an Asian
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2017-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hyun Joh, MD, PhD, Principal Investigator — East West Neo Medical Center
Locations (1):
- Vascular Surgery, Kyung Hee University East-West Neo Medical Center, Seoul, South Korea